CLINICAL TRIAL: NCT01662193
Title: Effects of Vitamin D and Calcium Supplementation on Inflammatory Biomarkers and Adypocytokines in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Marjan Tabesh, Director, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190136
Record Dates: First submitted 2012-07-29; First posted 2012-08-10 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Nutritional and Metabolic Disease
Keywords: Cholecalciferol; Calciol; vitamin D3; Diabetes Mellitus; Diabetes Mellitus Type 2; glucose metabolism disorders; ergocalciferol; calcium; adipicytokines; inflammatory biomarkers
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- vitamin D3 (Experimental): vitamin D3 supplement 50000 IU vitamin D3 per week
  Interventions: Dietary Supplement: vitamin D3 supplement
- calcium supplement (Experimental): calcium supplement 1000 mg calcium carbonate daily
  Interventions: Dietary Supplement: calcium supplement
- vitamin D and calcium supplement (Experimental): vitamin D3 and calcium supplementation 50000 IU vitamin D3 per week and 1000 mg calcium carbonate daily
  Interventions: Dietary Supplement: vitamin D3 and calcium supplement
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: vitamin D3 supplement
  Other Names: cholecalciferol
  Arms: vitamin D3
Dietary Supplement: calcium supplement
  Other Names: calcium carbonate
  Arms: calcium supplement
Dietary Supplement: vitamin D3 and calcium supplement
  Other Names: cholecalciferol and calcium carbonate
  Arms: vitamin D and calcium supplement
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
The epidemic of type 2 diabetes is an enormous public health problem in all parts of the world, with 366 million cases by 2030. Chronic inflammation has been postulated to play a role in the pathogenesis of type 2 diabetes. High levels of adiponectin and inflammatory biomarkers are known as a new risk factor for diabetes. There is accumulating evidence suggesting that altered vitamin D and calcium homeostasis affect the development of type 2 diabetes, but it is still unclear whether that effects are through reducing the level of adipocytokines and inflammatory biomarkers or not. This study has been designed to evaluate the effects of vitamin D and calcium supplementations alone and in combination on inflammatory biomarkers and adypocytokines in type 2 diabetic patients.

This study is a single masked, controlled randomized trial with period of 8 weeks. 120 diabetic patients who met the inclusion criteria will enroll in this study. Subjects will randomly assign in to four groups. Randomization will be achieved by permuted blocks with stratification by age, sex, BMI, type of diabetes and dose of medication. Group1 will receive 50000 IU of vitamin D3 per week plus calcium placebo, group2 will received 1000 mg of calcium carbonate per day plus vitamin D placebo, group 3 will receive 50000 IU of vitamin D3 plus 100 of mg calcium carbonate per day and group four will receive calcium and vitamin D placebos. Total cholesterol, HDL, LDL, serum triglyceride, serum glucose, serum insulin, HbA1C, leptin, adiponectin and inflammatory biomarkers such as TNF-alpha, IL-6 and high sensitivity C reactive protein (hs-CRP) will be determine by taking blood samples at the baseline and at the end of intervention. Systolic and diastolic blood pressure and anthropometric measurements (height, weight, hip and waist circumferences) will be measured at the baseline and after 8 weeks of intervention. 3 dietary records and 3 physical activity records will be taken at 2,4 and 6 week of intervention to make sure that all subjects maintain their usual diet and physical activity during intervention.

ELIGIBILITY:
Inclusion Criteria:

* more than 30 years old
* have no history of renal failure, cancer, liver diseases, thyroid diseases or any other inflammatory diseases
* have no allergy
* do not use any tobacco products
* not using corticosteroids
* not consuming any kinds of vitamin D or calcium supplement
* have not more than 4 kilograms weight change during last 3 months

Exclusion Criteria:

* pregnancy
* insulin dependent diabetes

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
change in inflammatory biomarkers from baseline at 8 weeks | 8 weeks
  including:IL-6, TNF-alpha, hs-CRP
change in adipocytokines from baseline at 8 weeks | 8 weeks
  including: adiponectin and leptin

SECONDARY OUTCOMES:
change in weight (Kg) from baseline at 8 weeks | 8 weeks
change in lipid profile from baseline at 8 weeks | 8 weeks
  including: LDL, HDL, total cholesterol, TG
change in serum Glucose from baseline at 8 weeks | 8 weeks
change in height (Cms) from baseline at 8 weeks | 8 weeks
change in hip circumference (Cms) from baseline at 8 weeks | 8 weeks
change in waist circumference (Cms) from baseline at 8 weeks | 8 weeks
change in serum Insulin from baseline at 8 weeks | 8 weeks
change in HbA1C from baseline at 8 weeks | 8 weeks
change in blood pressure from baseline at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School of Isfahan, Isfahan, Isfahan, Iran

REFERENCES:
- [Derived] Tabesh M, Azadbakht L, Faghihimani E, Tabesh M, Esmaillzadeh A. Effects of Calcium Plus Vitamin D Supplementation on Anthropometric Measurements and Blood Pressure in Vitamin D Insufficient People with Type 2 Diabetes: A Randomized Controlled Clinical Trial. J Am Coll Nutr. 2015;34(4):281-9. doi: 10.1080/07315724.2014.905761. Epub 2015 Mar 4. PMID 25738212
- [Derived] Tabesh M, Azadbakht L, Faghihimani E, Tabesh M, Esmaillzadeh A. Calcium-vitamin D cosupplementation influences circulating inflammatory biomarkers and adipocytokines in vitamin D-insufficient diabetics: a randomized controlled clinical trial. J Clin Endocrinol Metab. 2014 Dec;99(12):E2485-93. doi: 10.1210/jc.2014-1977. PMID 25215557
- [Derived] Tabesh M, Azadbakht L, Faghihimani E, Tabesh M, Esmaillzadeh A. Effects of calcium-vitamin D co-supplementation on metabolic profiles in vitamin D insufficient people with type 2 diabetes: a randomised controlled clinical trial. Diabetologia. 2014 Oct;57(10):2038-47. doi: 10.1007/s00125-014-3313-x. Epub 2014 Jul 10. PMID 25005333